CLINICAL TRIAL: NCT03041389
Title: A Computerized Cognitive Behavioral Therapy Randomized, Controlled, Pilot Trial for Insomnia in Parkinson Disease (The ACCORD-PD Study)
Brief Title: Computerized Cognitive Behavioral Therapy Trial for Insomnia in Parkinson Disease
Acronym: ACCORD-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Anwar Ahmed, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-1388
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Insomnia Related to Specified Disorder; Parkinson Disease
Keywords: Computerized Cognitive Behavioral Therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized (1:1 ratio), single-blind, parallel-group, controlled study
Who Masked: Outcomes Assessor
Masking Description: The rater of outcomes questionnaires is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCBT-I Group (Experimental): The patients who will be randomized to CCBT-I group will get Cleveland Clinic CCBT-I program through the internet (Cleveland Clinic Wellness Go! To Sleep six-week online program). The program involves a 6-week effective sleep therapy, an online sleep log and daily sleep score, six specially crafted relaxation practices, daily sleep improvement recommendations, activities to help the patient get the sleep needed, daily e-mails from the patient's program coach, daily articles to help the patient get the most out of the program and a mobile application for easy sleep tracking.
  Interventions: Behavioral: CCBT-I Group
- Control Group (Active Comparator): The patients who will be randomized control group will be given a reading material only including recommendations about sleep hygiene, stimulus control and sleep restriction. The control group will have access to the CCBT-I program through the internet (Cleveland Clinic Wellness Go! To Sleep six-week online program), if proven effective, after the study is completed.
  To identify PD-specific barriers to Internet usage and CCBT-I, all patients at the end of the study or at the time of drop out will have a questionnaire on the barriers to CCBT-I.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: CCBT-I Group — Every patient will have a unique password to access to CCBT-I. The program consists of 5 cores: sleep log, day's lesson, activities, relaxation and progress. Each day, the patients fill in sleep logs before getting the day's lesson. Filling sleep log will be reminded daily by the program coach from Sleep Center.
  Arms: CCBT-I Group
Behavioral: Control Group — Reading material only including recommendations about sleep hygiene, stimulus control and sleep restriction. Access to the CCBT-I program through the internet (Cleveland Clinic Wellness Go! To Sleep six-week online program), if proven effective, after the study is completed.
  Arms: Control Group

SUMMARY:
The therapeutic options are limited in Parkinson's Disease (PD) patients with insomnia and are often based on pharmacological treatments. It has been shown that the cognitive behavioral therapy can be effective in primary insomnia. To the investigators knowledge, the effect of computerized cognitive behavioural therapy on insomnia in PD has not been evaluated before. The aim of this study is to demonstrate the beneficial effects of 6-weeks of computerized cognitive behavioural therapy on clinical and sleep variables of insomnia in Parkinson's disease patients.

DETAILED DESCRIPTION:
The investigators propose a randomized (1:1 ratio), single-blind, parallel-group, controlled study on Computerized cognitive behavioral therapy for insomnia (CCBT-I) treatment for PD patients which evaluates clinical and sleep variables before and after 6-week CCBT-I.

28 subjects with idiopathic PD having insomnia will be recruited for this study. Insomnia will be defined by >11 Insomnia Severity Index (ISI) scores as 11 was found in a study examining sensitivity/specificity for ISI cutoffs to be highest % correctly identified in clinical sample.

After a screening visit, the patients will be randomized to either the CCBT-I 6-week treatment arm or the control treatment arm. At the end of the screening patients will also receive 2 enveloped packages of questionnaires to be completed at Week 8 and Week 12 (after baseline) at home and mailed back to the Principal Investigator (PI) at the study center. The patients will get a follow-up phone call every week for the treatment period and during Week 8 and Week 12 to remind them to complete evaluations and mail back to the PI.

The Cleveland Clinic Wellness Institute will also send weekly email prompts to the participants in the CCBT-I treatment arm to ensure/improve compliance with the online sleep program.

ELIGIBILITY:
Inclusion Criteria:

1. 35-85 years old PD patients, as diagnosed by a Movement Disorders neurologist
2. Male or Female
3. On the stable antiparkinsonian medication in the last 30 days
4. Having insomnia defined by >11 ISI scores
5. Access to a computer and internet
6. Be able to speak, read and understand English

Exclusion Criteria:

1. Dementia as defined by DSM-IV criteria
2. Patients with suboptimally treated depression and significant depressive symptoms as defined by a PHQ-9 score of >15 (PHQ-9 scores 1-4 Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression;20-27 Severe depression). Antidepressant medications, prescribed for depression or anxiety, will be allowed if the patient has been on a stable dose for at least 1 month.
3. Significant hallucinations or psychotic symptoms requiring antipsychotic medications
4. Presence of significant sleep disorders that could be contributing to insomnia such as known sleep apnea, PLMS, RBD, RLS on screening exam by medical history and neurological exam.
5. Presence of significant motor fluctuations, especially nocturnal akinesia that could be contributing to insomnia
6. Use of sedatives, benzodiazepines or sedating anti-depressants (such as mirtazapine, TCAs), modafinil, stimulants, anticholinergic medications, zolpidem, zopiclone, eszopiclone, zaleplon will be allowed if the the patient has been on a stable dose for at least 1 month and if not taken as a sleep aid.
7. Significant renal, hepatic, cardiac and thyroid disease that can interfere with protocol adherence

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | 12 weeks
  To demonstrate a significant difference in the mean Insomnia Severity Index (ISI), from baseline to Week 12 among subjects randomized to CCBT-I treatment versus the control group

SECONDARY OUTCOMES:
Pittsburgh Insomnia Rating Scale | 12 weeks
  To demonstrate a significant difference in the mean Pittsburgh Insomnia Rating Scale (PIRS-20) from baseline to Week 12 among subjects randomized to CCBT-I treatment versus the control group
Total Sleep Time | 12 weeks
  To demonstrate a significant increase in Total Sleep Time (TST) in PD subjects, from baseline to Week 12, who were randomized to CCBT-I via daily sleep logs in the online program as compared to the control group
Patient Global Impression of Improvement | 12 weeks
  To demonstrate a significant difference in the number of patients who significantly improved based on Patient Global Impression of Improvement (PGI-I) from baseline to Week 12 among subjects randomized to CCBT-I treatment versus the control group
Fatigue Severity Scale | 12 weeks
  To demonstrate a significant difference in the mean Fatigue Severity Scale (FSS), from baseline to Week 12 among subjects randomized to CCBT-I treatment versus the control group
Epworth Sleepiness Scale | 12 weeks
  To demonstrate a significant difference in the mean Epworth Sleepiness Scale (ESS), from baseline to Week 12 among subjects randomized to CCBT-I treatment versus the control group

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Ahmed, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No
No IPD made available to other researchers.